CLINICAL TRIAL: NCT03468101
Title: Characterization of Professional COPD Related to Exposure to Organic Dust - Mean Follow up at 6 Years
Acronym: BALISTIC 2
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: R/2016/53
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COPD; Exposure Occupational
Keywords: COPD; Dairy farmers; Exposure Occupational; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Physiological Phenomena; Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dairy farmers COPD
  Interventions: Other: Pulmonary Function Testing
- Non farmers COPD
  Interventions: Other: Pulmonary Function Testing

INTERVENTIONS:
Other: Pulmonary Function Testing — Pulmonary Function Testing, Cardiopulmonary exercise testing, 6 Minute walk test, Thoracic CT
  Other Names: Cardiopulmonary exercise testing; 6 Minute walk test; Thoracic CT

SUMMARY:
The main objective of the BALISTIC research program is to characterize COPD related to organic particles (of which the model is agricultural COPD) in comparison with tobacco-related COPD, at the clinical, functional (at rest and exercise), inflammatory and physiopathological level.

The cross-sectional step BALISTIC 1 made it possible to include 400 patients between 2011 and 2015, and to identify approximately 100 dairy farmers COPD and 100 non-dairy farmers COPD (tobacco COPD). Preliminary results, as well as those of an ancillary study that included a group of subjects exposed to mineral dust and fumes, suggest that agricultural COPD is a predominantly non-emphysematous or essentially bronchial disease with IgE-mediated allergic mechanisms.

The current project BALISTIC 2 proposes to conduct a comparative study at + 6 years on average of the two groups of COPD subjects identified in BALISTIC 1 in order to specify the phenotype of COPD in dairy farmers by, in particular, the study of the rate of decline of resting and exercise respiratory function parameters, its computed tomography presentation and its genetic and epigenetic profile.

The prospects of this work are to improve the management of COPD in any cause by setting up preventive and curative therapeutic approaches in order to provide answers to the progression of a disease that makes part of the few major public health problems of the 21st century.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated to BALISTIC 1 and who had been diagnosed with COPD, belonging to either the "dairy farmers COPD" group or the "non farmers COPD" group.

Exclusion Criteria:

-

Ages: 46 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who participated to BALISTIC 1 and who had been diagnosed with COPD, belonging to either the "dairy farmers COPD" group or the "non farmers COPD" group.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Annual change in FEV1 judged by two spirometry performed on average at 6-year intervals and expressed in ml per year. | two spirometry performed on average at 6-year
  Annual change in FEV1 judged by two spirometry performed on average at 6-year intervals and expressed in ml per year.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No